CLINICAL TRIAL: NCT00339612
Title: NISDI Pediatric Latin American Countries Epidemiologic Study (PLACES): A Prospective Observational Study of HIV-Infected Children at Clinical Sites in Latin American Countries
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902270; 02-CH-N270
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: HIV
Keywords: Perinatal; HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HIV-infected children who acquired HIV infection through mothe: HIV-infected children in who acquired HIV infection through mother-to-child transmission (MTCT).

SUMMARY:
This is an observational, prospective cohort study to describe the demographic, clinical, immunologic, and virologic characteristics of HIV-infected children at participating clinical sites in Latin American countries. Enrollment in this study will consist of approximately 500 HIV-infected children in two cohorts who acquired HIV infection through mother-to-child transmission (MTCT). The first group will be a static cohort consisting of HIV-infected children who were five years of age or younger when previously enrolled into the NISDI Pediatric Protocol. The second cohort will be a dynamic cohort of prospectively enrolled, HIV-infected children who are five years of age or younger. We will characterize complications from both the disease and its treatments. Subjects will be evaluated every six months for approximately five years and assessments of growth, morbidity, disease progression and mortality will be made.

DETAILED DESCRIPTION:
This is an observational, prospective cohort study to describe the demographic, clinical, immunologic, and virologic characteristics of HIV-infected children at participating clinical sites in Latin American countries. Enrollment in this study will consist of approximately 500 HIV-infected children in two cohorts who acquired HIV infection through mother-to-child transmission (MTCT). The first group will be a static cohort consisting of HIV-infected children who were five years of age or younger when previously enrolled into the NISDI Pediatric Protocol. The second cohort will be a dynamic cohort of prospectively enrolled, HIV-infected children who are five years of age or younger. We will characterize complications from both the disease and its treatments. Subjects will be evaluated every six months for approximately five years and assessments of growth, morbidity, disease progression and mortality will be made.

ELIGIBILITY:
* INCLUSION CRITERIA:

Static Cohort:

1. Previous participation in a NISDI Protocol
2. Less then 6 years of age (before their 6th birthday) at the time of enrollment into the NISDI Pediatric Protocol
3. HIV-infected
4. HIV infection must be documented in the medical records by:

   1. For children less than 18 months old when tested, two or more of the following (separate determinations on separate blood specimens):

      * Positive HIV culture
      * Positive HIV DNA PCR
      * Positive neutralizable p24 antigen
      * Quantitative HIV RNA greater than or equal to 10,000 copies/ml
   2. For children greater than or equal to 18 months old when tested, two or more of the following (separate determinations on separate blood specimens):

      * Reactive test for HIV antibody in a sample obtained at greater than or equal to 15 months of age with confirmatory test by Western Blot or Immunofluorescence assay
      * Positive HIV culture
      * Positive HIV DNA PCR
      * Positive neutralizable p24 antigen
      * Quantitative HIV RNA greater than or equal to 1,000 copies/ml
5. Documentation of maternal HIV infection by country appropriate National Guidelines
6. Signed informed consent from parent or legal guardian. An informed assent document will be provided for children 8 years of age or older when appropriate.
7. Subjects must be able to be followed at a participating clinical site.
8. Subjects may be co-enrolled in clinical trials for treatment of HIV infection, opportunistic infections, or other HIV-related effects.

Dynamic cohort:

1. HIV-infected less then 6 years of age (before their 6th birthday) at enrollment into this protocol
2. HIV infection documented by:

   1. For children <18 months old when tested, two or more of the following (separate determinations on separate blood specimens):

      * Positive HIV culture
      * Positive HIV DNA PCR
      * Positive neutralizable p24 antigen
      * Quantitative HIV RNA greater than or equal to 10,000 copies/ml
   2. For children greater than or equal to 18 months old when tested, two or more of the following (separate determinations on separate blood specimens):

      * Reactive test for HIV antibody in a sample obtained at greater than or equal to 15 months of age with confirmatory test by Western Blot or Immunofluorescence assay
      * Positive HIV culture
      * Positive HIV DNA PCR
      * Positive neutralizable p24 antigen
      * Quantitative HIV RNA greater than or equal to 1,000 copies/ml
3. Documentation of maternal HIV infection by country appropriate National Guidelines
4. Signed informed consent from parent or legal guardian. An informed assent document will be provided for children 8 years of age or older when appropriate.
5. Subjects must be able to be followed at a participating clinical site
6. Subjects may be co enrolled in clinical trials for treatment of HIV infection, opportunistic infections, or other HIV related effects

EXCLUSION CRITERIA:

1. Children who are born to an HIV infected mother, but are uninfected or of indeterminate HIV infection status
2. Children who are orphans without legal guardians or are wards of the state

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 500 HIV-infected children in two cohorts who acquired HIV infection through mother-to-child transmission (MTCT). The first group will be a static cohort consisting of HIV-infected children who were five years of age or younger when previously enrolled into the NISDI Pediatric Protocol. The second cohort will be a dynamic cohort of prospectively enrolled, HIV-infected children who are five years of age or younger. We will characterize complications from both the disease and its treatments. Subjects will be evaluated every six months for approximately five years and assessments of growth, morbidity, disease progression and mortality will be made.
Sampling Method: Non-Probability Sample
Enrollment: 2129 (Actual)
Dates: Start 2002-07-30 (Actual); Primary Completion 2011-12-30 (Actual); Study Completion 2020-07-28 (Actual)

SECONDARY OUTCOMES:
HIV RNA copies | q 6 months
  characterize complications from both the disease and its treatments
CD4 + T cell count | q 6 months
  characterize complications from both the disease and its treatments
medical history | q 6 months
  characterize complications from both the disease and its treatments
hematology and chemistry labs | q 6 months
  characterize complications from both the disease and its treatments

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Hazra, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (14):
- Brazil (12):
  - Universidade Federal de Minas Gerais, Belo Horizonte
  - Ricardo de Souza STD/HIV Clinic-Caxias do Sul, Caxias do Sul
  - Hospital Conceicao, Porto Alegre
  - Hospital de Clinicas, Porto Alegre
  - Hospital Femina, Porto Alegre
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital dos Servidores do Estado, Rio de Janeiro
  - Hospital Geral Nova de Iguacu, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagao Gesteira, Rio de Janeiro
  - Federal University of Sao Paulo-Escola Paulista de Medicina, São Paulo
  - Hospital das Clinicas da Falculdade De Medinica, São Paulo
  - Instituto de Infectologica Emilio Ribas (IIER), São Paulo
- Hospital Infantil de Mexico Federico Gomez (HIM), Mexico City, Mexico
- University of San Marcos, Lima, Peru

REFERENCES:
- [Background] Connor EM, Sperling RS, Gelber R, Kiselev P, Scott G, O'Sullivan MJ, VanDyke R, Bey M, Shearer W, Jacobson RL, et al. Reduction of maternal-infant transmission of human immunodeficiency virus type 1 with zidovudine treatment. Pediatric AIDS Clinical Trials Group Protocol 076 Study Group. N Engl J Med. 1994 Nov 3;331(18):1173-80. doi: 10.1056/NEJM199411033311801. PMID 7935654
- [Background] Wade NA, Birkhead GS, Warren BL, Charbonneau TT, French PT, Wang L, Baum JB, Tesoriero JM, Savicki R. Abbreviated regimens of zidovudine prophylaxis and perinatal transmission of the human immunodeficiency virus. N Engl J Med. 1998 Nov 12;339(20):1409-14. doi: 10.1056/NEJM199811123392001. PMID 9811915
- [Background] Lindegren ML, Byers RH Jr, Thomas P, Davis SF, Caldwell B, Rogers M, Gwinn M, Ward JW, Fleming PL. Trends in perinatal transmission of HIV/AIDS in the United States. JAMA. 1999 Aug 11;282(6):531-8. doi: 10.1001/jama.282.6.531. PMID 10450714